CLINICAL TRIAL: NCT01017614
Title: A Phase III, Randomized, Comparative, Open-label Study of Intravenous Iron Oligosaccharide (Monofer®) Administered by Infusions or Repeated Bolus Injections in Comparison With Oral Iron Sulphate in Inflammatory Bowel Disease Subjects With Iron Deficiency Anaemia
Brief Title: Iron Oligosaccharide in Inflammatory Bowel Disease Subjects With Iron Deficiency Anaemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmacosmos A/S (Industry)
Collaborators: Max Neeman International (Unknown)
Responsible Party: Vice President, Clinical Development, Pharmacosmos A/S
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P-Monofer-IBD-01; EudraCT no 2009-012544-16
Record Dates: First submitted 2009-11-19; First posted 2009-11-20 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Inflammatory Bowel Disease
Keywords: Inflammatory Bowel Disease; Iron deficiency; Iron deficiency anaemia; Anaemia
MeSH Terms: conditions — Inflammatory Bowel Diseases; Iron Deficiencies; Anemia, Iron-Deficiency; Anemia | interventions — Iron-Dextran Complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monofer (Experimental): * administered as intravenous infusions (A1)
  * administered as intravenous bolus injections (A2)
  Interventions: Drug: Monofer
- Iron Sulphate (Active Comparator): tablets administered orally
  Interventions: Drug: Iron Sulphate

INTERVENTIONS:
Drug: Monofer — * administered as intravenous infusions (A1)repeated weekly until total iron repletion is obtained
  * administered as intravenous bolus injections (A2)as repeated bolus injections weekly until total iron repletion is obtained
  Arms: Monofer
Drug: Iron Sulphate — 200 mg daily
  Arms: Iron Sulphate

SUMMARY:
The purpose of the trial is to demonstrate that intravenous iron oligosaccharide is non-inferior to oral iron sulphate in reducing iron deficiency anaemia secondary to inflammatory bowel disease (IBD), evaluated as the ability to increase haemoglobin (Hb).

DETAILED DESCRIPTION:
The study is designed to determine the effects of an investigational drug Monofer in subjects with Inflammatory Bowel Disease (IBD) (an intestinal disease characterized by swelling, redness and sometimes ulcers in intestine) and with Iron Deficiency Anaemia (IDA) (Anaemia is a condition characterized by deficiency of blood in the body).

ELIGIBILITY:
Inclusion Criteria:

Subjects with a diagnosis of IBD with iron deficiency anaemia will be included if they meet all of the following criteria:

1. Men and women, aged more than 18 years.
2. Subjects diagnosed with inflammatory bowel disease and mild to moderate disease activity (defined as a score of less than or equal to 5 on the Harvey-Bradshaw index for Crohn's disease and a Mayo score (subscore without endoscopy) of less than or equal to 6 for ulcerative colitis).
3. Hb <12.0 g/dL (7.45 mmol/L).
4. Transferrin saturation (TfS) <20 %.

Exclusion Criteria:

1. Anaemia predominantly caused by other factors than iron deficiency anaemia.
2. Iron overload or disturbances in utilisation of iron (e.g. haemochromatosis and haemosiderosis).
3. Drug hypersensitivity (i.e. previous hypersensitivity to Iron Dextran or iron mono- or disaccharide complexes or to iron sulphate).
4. Known hypersensitivity to any excipients in the investigational drug products.
5. Subjects with a history of multiple allergies.
6. Active Intestinal Tuberculosis.
7. Active Intestinal amoebic infections.
8. Decompensated liver cirrhosis and hepatitis (alanine aminotransferase (ALT) > 3 times upper limit normal).
9. Acute infections (assessed by clinical judgement), supplied with white blood cells (WBC) and C-reactive protein (CRP)).
10. Rheumatoid arthritis with symptoms or signs of active joint inflammation.
11. Pregnancy and nursing
12. Extensive active bleeding necessitating blood transfusion.
13. Planned elective surgery during the study.
14. Participation in any other clinical study within 3 months prior to screening.
15. Intolerance to oral iron treatment.
16. Untreated B12 or folate deficiency.
17. Other I.V. or oral iron treatment or blood transfusion within 4 weeks prior to screening visit.
18. Erythropoetin treatment within 8 weeks prior to screening visit.
19. Diagnosis of Hepatitis B and/or C, confirmed by appropriate lab test.
20. Any other medical condition that, in the opinion of Investigator, may cause the patient to be unsuitable for the completion of the study or place the patient at potential risk from being in the study. Example, Uncontrolled Hypertension, Unstable Ischemic Heart Disease or Uncontrolled Diabetes Mellitus.
21. History of immunocompromise, including positive HIV test result

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2009-10; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Change in Hb concentration from baseline to week 8. | 8 weeks

SECONDARY OUTCOMES:
Number of subjects who achieve target limits of Hb (men 13-18 g/dL, women 12-16 g/dL) and have change in Hb concentration > 1.0 g/dL and have serum ferritin (100-800µg/L) and have achieved Transferrin saturation (TfS) (20-50 %) at week 2, 4 and 8. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pharmacosmos A/S, Study Chair — Pharmacosmos A/S, Roervangsvej 30, DK 4300 Holbaek, Denemark
Locations (10):
- Denmark (3):
  - Research Site, Aalborg
  - Research Site, Aarhus
  - Research Site, Copenhagen
- India (6):
  - Research Site, Hyderabad
  - Research Site, Jaipur
  - Research Site, Mumbai
  - Research Site, Nashik
  - Research Site, New Delhi
  - Research Site, Pune
- Research Site, London, United Kingdom